CLINICAL TRIAL: NCT07298122
Title: Cardiac Assessment for Thrombus Detection in the Heart Using Advanced Imaging (MRI, CT) in ESUS With Left Ventricular Disease
Acronym: CATCH ME
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 5684
Record Dates: First submitted 2025-12-11; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cryptogenic Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Embolic stroke of undetermined source with left ventricular disease: Patients with embolic stroke of undetermined source and left ventricular disease, with no intracardiac thrombus identified on transthoracic echocardiography, will undergo advanced cardiac imaging such as cardiac MRI and/or CT

SUMMARY:
The CATCH ME study is a prospective, multicenter, observational, no-profit study aimed at improving embolic risk stratification in patients with embolic stroke of undetermined source (ESUS), particularly in those with left ventricular disease (LVD). LVD is defined by a mildly to moderately reduced ejection fraction (30-49%), left ventricular wall motion abnormalities (hypo/akinesia), ventricular dilation, cardiomyopathies, and other related conditions. In these patients, the intermittent formation of intracardiac thrombi within the ventricle, often undetectable by standard diagnostic evaluation such as transthoracic echocardiography (TTE) alone, may serve as an unrecognized embolic source. However, in clinical practice, such patients are frequently discharged on antiplatelet therapy alone, without adequate thromboembolic risk stratification, thus leaving them at a high risk of ischemic recurrence. This study aims to assess the additional diagnostic value of advanced cardiac imaging - Cardiac Magnetic Resonance Imaging (CMRI) and/or Cardiac Computed Tomography (CCT) - in detecting intracardiac thrombi not identified by TTE in patients with ESUS and LVD.

DETAILED DESCRIPTION:
ESUS is a subgroup of ischemic stroke characterized by several potential embolic sources and represents a significant challenge in clinical management. Among ESUS patients, those with LVD, defined as a mildly to moderately reduced ejection fraction (30-49%), left ventricular wall motion abnormalities (LVWMAs), ventricular dilation, cardiomyopathies, and other related conditions, constitute a high-risk subgroup for adverse outcomes. In this population, the underlying stroke mechanism could be the intermittent formation of intraventricular thrombi. Factors such as low cardiac output, dilated cardiac chambers, poor contractility, and endothelial dysfunction may activate Virchow's triad, thereby increasing the risk of thrombosis. The standard cardiac diagnostic approach for these patients typically includes TTE, which is often unable to detect small intracardiac thrombi, due to their transient nature or the limited sensitivity of TTE. This limitation may lead to a diagnostic gap, with the potential risk of not implementing adequate secondary prevention therapy. In fact, these patients are usually discharged with antiplatelet therapy, despite several studies showing a higher risk of stroke recurrence. Advanced cardiac imaging techniques, including CCT and CMRI, are increasingly being used in the diagnostic evaluation of ESUS patients. Studies have demonstrated their role in identifying significant vascular and cardiac abnormalities not otherwise detected by TTE, leading to a reclassification of the stroke etiology and a consequent reduction in the ESUS prevalence. Current AHA/ASA guidelines recommend the use of advanced cardiac imaging (CMRI and CCT) in selected ESUS cases to optimize preventive therapy and reduce the risk of recurrence (class 2b, level of evidence C). CMRI, in particular, is recommended when (1) there is suspicion of an intracardiac thrombus but TTE results are inconclusive, or (2) TTE is negative but there remains a clinical suspicion of a cardioembolic stroke etiology. Studies have shown that both CCT and CMRI allow for the detection of cardiac thrombi significantly more often than TTE in ESUS patients, especially those with markers of LVD. CMRI is considered the gold standard for non-invasive evaluation of the left ventricle and has the highest sensitivity in detecting ventricular thrombi. Despite the relatively widespread use of advanced cardiac imaging in selected ESUS cases, there is currently a lack of systematic data on its clinical utility in this specific population. This study aims to assess the role of advanced cardiac imaging (CMRI and/or CCT) in detecting intracardiac thrombi in ESUS patients with LVD compared to the use of TTE alone. This study intends to provide real-world evidence on the additional diagnostic value of advanced cardiac imaging, contributing to a better understanding of its utility in secondary stroke prevention.

The study will last for three years, with a recruitment period of two years and 1 year of follow-up. It will be conducted in three phases:

1. Initial Screening Phase (Phase 1): Inclusion of all ESUS patients with acute ischemic stroke and LVD. Patients with thrombi detected via TTE will be classified as cardioembolic and excluded from the ESUS subgroup analysis, but included in the initial data collection phase to assess the prevalence of ventricular thrombi in this population.
2. Imaging Phase (Phase 2): This phase will focus on the subgroup of patients classified as ESUS with LVD, where no thrombi were detected by TTE, and who will undergo advanced cardiac imaging (CMRI, CCT), as recommended by current guidelines, within 15 days from the index ischemic event.
3. Follow-up (Phase 3): All recruited patients (both those classified as cardioembolic and ESUS) will be followed for a period of 24 months to monitor the occurrence of vascular events, recurrent ischemic stroke, hemorrhagic events, atrial fibrillation, mortality, and any therapeutic modifications.

The main goal is to evaluate the diagnostic effectiveness of advanced cardiac imaging (CMRI and/or CCT) in identifying intracardiac thrombi in ESUS patients with LVD who have negative TTE results (no thrombi). The study will also aim to determine the prevalence of intracardiac thrombi detected by TTE in all patients with ESUS and LVD. Additionally, it will assess the clinical and cardiac differences between patients based on whether thrombi are present and the method used for detecting them. The study will examine how the results from CMRI and/or CCT influence therapeutic decisions, such as the initiation of anticoagulant therapy when thrombi are found. Furthermore, the study will evaluate the risk of adverse events during follow-up, including recurrent strokes, coronary events, major bleeding episodes, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years Modified Rankin Scale (mRS) score ≤ 4 Diagnosis of acute ischemic stroke (detected by CT or brain MRI) Diagnosis of ESUS according to standard criteria
* Stroke detected by CT or MRI that is not lacunar. Lacunar is defined as a subcortical infarction (including pons and mesencephalon) in the distribution of the small penetrating cerebral arteries, with a maximum size ≤ 1.5 cm on CT or ≤ 2.0 cm on diffusion-weighted MRI images (< 1.5 cm on T2-weighted MRI images). Excluded: multiple small deep infarcts, lateral bulb infarcts, cerebellar infarcts, patients with clinical lacunar stroke syndrome and no visible infarction on imaging.
* Absence of extracranial or intracranial atherosclerosis causing ≥ 50% stenosis in the artery supplying the ischemic area. Vascular imaging of the extracranial and intracranial vessels is required using angiography, CT angiography (CTA), MR angiography (MRA), or color Doppler ultrasound, at the discretion of the treating physician and local principal investigator.
* No major cardioembolic source identified, including permanent or paroxysmal atrial fibrillation (AF), sustained atrial flutter, intracardiac thrombus (*as specified above, these patients will be recruited in phase 1 of the study only if an isolated ventricular thrombus is found without other major cardiac causes), mechanical heart valve prosthesis, atrial myxoma or other cardiac tumors, moderate or severe mitral stenosis, recent myocardial infarction (< 4 weeks), left ventricular ejection fraction (EF) < 30%, valve vegetations or infective endocarditis.
* No other identified cause of stroke (such as arteritis, dissection, migraine, vasospasm, drug abuse, hypercoagulability, etc.)

Presence of LVD defined by at least one of the following criteria:

* Moderately reduced left ventricular (LV) systolic function, defined as EF 30-49%.
* LV wall motion abnormalities (LVWMAs), defined as hypokinetic, akinetic, or dyskinetic segments of the left ventricular wall not associated with recent or acute myocardial infarction (within 4 weeks).
* LV aneurysm
* Enlarged LV with or without spontaneous contrast
* Non-compacted LV, with deep trabeculations or spongy LV
* Cardiomyopathies, such as restrictive cardiomyopathy, hypertrophic cardiomyopathy, or cardiac amyloidosis

Patients capable of signing informed consent (IC) or, in the case of unconscious patients without an authorized legal representative, recruited in a "Deferred" mode

Exclusion Criteria:

* Major cardioembolic sources, as specified in the ESUS criteria Patients with a thrombophilic state secondary to active cancer, defined as "diagnosis of solid or hematologic malignant tumor within 6 months of stroke, ongoing oncological treatment, or hematologic cancer not in remission." Patients with ipsilateral carotid plaques to the ischemic stroke considered at high risk: thrombus on the wall, floating thrombus, ulcerated plaque.

Patients under 60 years of age with a high-risk patent foramen ovale (PFO) and stroke classified as "probable" PFO-associated stroke according to the PASCAL classification.

Pregnancy or puerperium. Contraindication to MRI and CT with contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 85 years, with an mRS score ≤ 4 and Ischemic stroke classified as ESUS according to standard criteria, with LVD (defined as moderately reduced ejection fraction 30-49%, presence of LC wall motion abnormalities, LV aneurysm, LV dilatation with or without spontaneous echo-contrast, non-compacted LV [with deep trabeculations or spongy LV], cardiomyopathies [severe restrictive cardiomyopathy, cardiac amyloidosis, hypertrophic cardiomyopathy]), in whom no intracardiac thrombi are identified on transthoracic echocardiogram and who are able to undergo advanced cardiac imaging (CMRI and/or CCT).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of left ventricular thrombus on advanced cardiac imaging (CMRI and/or CCT) | 15 days from the index stroke
  Prevalence of left ventricular thrombus detected by advanced cardiac imaging (CMR, CCT) compared with transthoracic echocardiography (TTE) in patients who underwent both investigations within 15 days of the index stroke

SECONDARY OUTCOMES:
Intracardiac thrombi detected by transthoracic echocardiography in all patients with ESUS and LVD. Recurrent ischemic stroke Systemic embolism Acute coronary events Major bleeding, defined by the International Society of Thrombosis and Hemostasis Mortal | 12 months from the index stroke
  Incidence of major cardiovascular events (MACE) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Cascio Rizzo, MD, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy, Italy